CLINICAL TRIAL: NCT03147937
Title: Assessing Postoperative Cognitive Changes After Major Joint Arthroplasty: A Prospective Cohort Study
Brief Title: Cognitive Changes After Major Joint Replacement - Full Trial (Cognigram 2)
Status: Active, not recruiting | Type: Observational
Sponsor: Dr. Stephen Choi (Other)
Responsible Party: Sponsor-Investigator, Dr. Stephen Choi, MD, FRCPC, MSc, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: 040-2017
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Cognitive Dysfunction; Cognitive Impairment; Mild Cognitive Impairment; Delirium; Cognitive Decline; Cognitive Change; Working Memory; Autoimmune Diseases; Inflammation
MeSH Terms: conditions — Postoperative Cognitive Complications; Cognitive Dysfunction; Delirium; Autoimmune Diseases; Inflammation | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cognitive Testing — Computerized CogState Brief Battery (CBB), Cognigram, assesses changes in four cognitive domains including psychomotor function, attention, learning and memory, and working memory. The CBB is a computerized test based on card games that can be administered online

SUMMARY:
Patients assume that cognitive performance rapidly returns to baseline after anesthesia and surgery. Several studies have shown that one week after major non-cardiac surgery about 27% of patients have postoperative cognitive dysfunction (POCD) and 10% of patients at 3 months. Very few studies have assessed the incidence of POCD beyond 3 months. POCD significantly reduces quality of life. Identifying risk factors for POCD is important because it is associated with prolonged hospital stay, loss of independence, and premature retirement. There is an urgent need to measure and document the level of cognitive change associated with surgery with an easy to use tool, both prior to admission and after discharge. This information can be used to plan appropriate care paths and to identify or test the efficacy of potential new treatments to alter the negative trajectory.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is thought to affect a significant proportion of patients after major surgery (up to 10% at 3 months). This is potentially a major public health issue because patients with POCD have prolonged hospital admission, loss of independence and mortality. Undoubtedly, if POCD is as prevalent and devastating as has been previously reported, the decision to undergo elective surgery should be influenced by the risk of developing POCD. Given the scope of the issue, the deficiencies in the literature surrounding POCD are concerning. There are many methodological issues with previous studies and the diagnosis of POCD in the perioperative period.

It is imperative that the true natures of postoperative cognitive changes are elucidated so that preoperative risk stratification can be appropriately determined. This will lead to care pathways and interventions that can modify any possible downward changes thereby reducing the negative impact on patients and the health care system.

Main Study Hypothesis: The incidence of postoperative cognitive changes in the joint arthroplasty population is influenced by:

1. Occurrence of major acute postoperative complications (e.g., cardiac event, pulmonary embolus, renal failure, pneumonia, prosthetic joint infection)
2. Pre-existing mild cognitive impairment (MCI)
3. Post-operative delirium
4. Pre-existing comorbid conditions with inflammatory states such as auto-immune disorders, coronary artery disease, obstructive sleep apnea, and auto-immune disorders

Study Objectives:

In patients undergoing primary total hip or knee arthroplasty the goals of this project are to:

1. Establish cognitive trajectories after major lower extremity joint arthroplasty and the incidence of both post-operative delirium and POCD
2. Test Main Study Hypothesis (see above)

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 50 years of age undergoing elective total hip or knee arthroplasty at Sunnybrook Health Sciences Centre

Exclusion Criteria:

* Lack of informed consent
* Inability to comply with study procedures or follow-up visits
* Patients with diagnosed dementia or those being treated with donepezil (Aricept®)
* Patients with severe cognitive impairment defined as baseline with a CBB score of equal to or less than 80 in at least one of the 4 CBB domains
* Patients with uncontrolled psychiatric diagnoses including schizophrenia, bipolar disorder, major depressive mood disorder
* Patients undergoing a second joint replacement & previously enrolled in this study within the past 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total hip arthroplasty (THA) or total knee arthroplasty (TKA) at the Holland Orthopedic and Arthritic Centre (HOAC) at Sunnybrook Health Sciences Centre (SHSC).
Sampling Method: Non-Probability Sample
Enrollment: 505 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Cognigram score decreasing by > 2 SDs from baseline at 4.5 | 4.5 months from baseline
  Proportion of patients with Cognigram score decreasing by > 2 SDs from baseline at 4.5

SECONDARY OUTCOMES:
Proportion of patients with Cognigram score decreasing between 1 and 2 standard deviations from baseline at 4.5 months | 4.5 months from baseline
  Proportion of patients with Cognigram score decreasing between 1 and 2 standard deviations from baseline at 4.5 months
Effect of pre-operative MCI on postoperative cognitive changes at 4.5 months | 4.5 months from baseline
  Effect of pre-operative MCI on postoperative cognitive changes at 4.5 months
Effect of pre-operative chronic inflammatory states on postoperative cognitive changes at 4.5 months | 4.5 months from baseline
  Effect of pre-operative chronic inflammatory states on postoperative cognitive changes at 4.5 months
Effect of postoperative delirium on postoperative cognitive changes at 4.5 months | 4.5 months from baseline
  Effect of postoperative delirium on postoperative cognitive changes at 4.5 months
Effect of postoperative complications on postoperative cognitive changes at 4.5 months | 4.5 months from baseline
  Effect of postoperative complications on postoperative cognitive changes at 4.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Choi, MD,FRCPC,MSc, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi S, Avramescu S, Orser BA, Au S. Protocol for a prospective cohort study of assessing postoperative cognitive changes after total hip and knee arthroplasty in the Greater Toronto area. BMJ Open. 2019 Feb 24;9(2):e024259. doi: 10.1136/bmjopen-2018-024259. PMID 30804030